CLINICAL TRIAL: NCT01136109
Title: A Prospective Pilot Study to Evaluate the Effect of Mechanical Ventilation on the Inferior Vena Cava Collapsibility Index
Brief Title: A Study to Evaluate the Effect of Mechanical Ventilation on the Inferior Vena Cava Collapsibility Index
Acronym: IVCCI
Status: Completed | Type: Observational
Sponsor: Naeem Ali, MD (Other)
Responsible Party: Sponsor-Investigator, Naeem Ali, MD, Associate Professor-Clinical, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2009H0143
Record Dates: First submitted 2010-05-26; First posted 2010-06-03 (Estimated); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Bedside ultrasound only: Bedside ultrasound to determine the dimensions of the inferior vena cava
- Ultrasound with ventilator changes: Bedside ultrasound to determine the dimensions of the inferior vena cava pre and post ventilator changes.

SUMMARY:
Previous research has shown that the Inferior Vena Cava Collapsibility Index (IVCCI) can be used to assess volume status. One limitation of the previous work is that changes in intra-thoracic pressure can influence this measurement, and the magnitude of this effect has never been described. The investigators aim is to correlate the degree of change in IVCCI with the set degree of change in intra-thoracic pressure in a heterogeneous population of critically ill patients.

DETAILED DESCRIPTION:
Initially eligible patients will be those admitted to the OSU MICU and 8ICU within the prior 48 hours. These patients will be screened for predetermined exclusion criteria. Eligible patients will have their IVCCI measured and baseline peak and plateau pressures noted. For those patients meeting a second set of criteria, a common ventilator maneuver will be preformed. The positive end-expiratory pressure will be increased by 5-10 cm/H20 pressure. This procedure will be aborted if ANY safety criteria are exceeded. During the interval, the IVCCI will be re-measured, the ventilator settings will be recorded, and the ventilator will be return to the initial settings. Since changes of these same magnitude are made daily in clinical practice, the risks to the patients in this study will be minimal and no more than that experienced in the course of usual care.

ELIGIBILITY:
Inclusion Criteria:

1. Age>17 years
2. Current use of mechanical ventilation through an endotracheal tube.
3. Admitted to ICU within last 48 hours

Exclusion Criteria:

1. Severe COPD by history (documented FEV1<50% predicted or CT evidence of emphysema)
2. Current suspected Asthma Exacerbation
3. Profound Hypoxia defined as a FiO2 requirement >90% or a PEEP >10 mmHg
4. Patient-ventilator desynchrony or active agitation
5. Unstable O2 requirement as determined by the primary clinical team.
6. Prisoners
7. Bedside clinician refusal (physician or treating nurse).

Exclusion Criteria for ventilator changes:

1. Cardiovascular instability (any increase in rate of vasopressors or i.v. fluid bolus for hypotension within the last four hours)
2. Current PEEP requirements of >15cmH2O
3. Current SpO2 of <88%.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: InpatientSample
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2009-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Determine the effect of an increase in positive end-expiratory pressure on intrathoracic pressure variables in patients with acute respiratory failure. | 24 months
  1. Determine the effect on inferior vena cava collapsibility index of an increase in positive end-expiratory pressure (and resultant change in mean airway pressure) in patients with acute respiratory failure.
  2. Determine the effect on central venous pressure of an increase in positive end-expiratory pressure (and resultant change in mean airway pressure) in patients with acute respiratory failure.
  3. Determine the effect on mean airway pressure of an increase in positive end-expiratory pressure in patients with acute respiratory failure.

SECONDARY OUTCOMES:
Determine the inter-rater reliability in obtaining inferior vena cava collapsibility index ultrasound images. | 24 months
Determine the relationship between central venous pressure and inferior vena cava collapsibility index at varying levels of mean airway pressure (MAP). | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Naeem Ali, M.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States